CLINICAL TRIAL: NCT05944315
Title: Introducing A Replicable Model For Injury Prevention Education In Kindergarten And First Grade Students
Brief Title: Injury Prevention Model For K-1 Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Good Samaritan Hospital Medical Center, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GoodSamaritanNY
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Trauma Injury; Child Behavior
Keywords: injury prevention; education model; elementary school children
MeSH Terms: conditions — Accidental Injuries; Child Behavior

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Participant
Masking Description: injury prevention knowledge being assessed in comparison to control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Teddy Bear Injury Prevention Clinic (Experimental): receiving injury prevention education
  Interventions: Behavioral: Education session
- Teddy Bear Hospital Education Clinic (Active Comparator): receiving hospital based education
  Interventions: Behavioral: Education session

INTERVENTIONS:
Behavioral: Education session — Classroom Education session appropriate for elementary school children

SUMMARY:
There is no educational injury prevention model uniquely suited for kindergarten and first grade (K-1) students. The Teddy Bear Injury Clinic (TBIC) is a unique modification of the teddy bear clinic to facilitate classroom injury prevention teaching

The TBIC will be administered to K-1 students, aged 5-7 years. Initial analysis will be descriptive and qualitative. Subsequent randomization of students to test and control groups followed by statistical analysis will be done to evaluate for effectiveness of the educational model

DETAILED DESCRIPTION:
The TBIC is a 40minute educational intervention divided into two sections with the first section consisting of classroom teaching with two safety messages each for four safety topics and the second section being that of students acting as caregivers for their teddy bears, using role-play for the messages taught.

Qualitative data collection will be initially done in an inductive manner and qualitative content analysis done using the directed method to analyze effectiveness and appropriateness of the TBIC for a pilot group.

Controlled trial will consist of randomizing students to either the TBIC group or the control group which will receive an alternate teddy bear clinic for non trauma related hospital education. Pre and post questionnaires will be administered to evaluate the efficacy of the TBIC.

Statistical analysis will be done using the Wilcoxon signed test rank score for the Likert scale based evaluations generated.

ELIGIBILITY:
Inclusion Criteria:

* K-1 elementary school students in the catchment area of the hospital for educational sessions

Exclusion Criteria:

* No consent/assent for study

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of Teddy Bear Injury Clinic for K-1 Students | 1 year
  Effectiveness of Teddy Bear Injury Clinic for K-1 Students for Injury Prevention Education

CONTACTS AND LOCATIONS:
Overall Officials: Vinci Jones, MD, Principal Investigator — Good Samaritan Hospital
Locations (1):
- Good Samaritan Hospital, West Islip, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Limited de-identified data and limited study details as specified below
Supporting Information: Study Protocol, SAP, ICF
Time Frame: for 1 year after study termination
Access Criteria: write to investigators with description of information necessary and reason for request

REFERENCES:
- [Result] Bloch YH, Toker A. Doctor, is my teddy bear okay? The "Teddy Bear Hospital" as a method to reduce children's fear of hospitalization. Isr Med Assoc J. 2008 Aug-Sep;10(8-9):597-9. PMID 18847160
- [Result] Kis H, Endres K, Karwowska A, Harrison M, Lau S, Lemire O, Zucker M. "Teddy Bear Hospital Project" school visits improve pre-clerkship students' comfort explaining medical concepts to children. Can Med Educ J. 2022 Jul 6;13(3):70-74. doi: 10.36834/cmej.73167. eCollection 2022 Jul. PMID 35875438